CLINICAL TRIAL: NCT06704789
Title: Investigation of the Possibility of Determining Cerebrovascular Disease Based on Hemodynamic Information of Localized Brain Regions
Status: Not yet recruiting | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Other Study IDs: 11-2024-059
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: EEG; FNIRS; Stroke; Normal
MeSH Terms: conditions — Stroke | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Hemorrhage stroke patients
  Interventions: Device: Measurement of brain activity (fNIRS, EEG)
- Ischemic stroke patients
  Interventions: Device: Measurement of brain activity (fNIRS, EEG)
- Healthy adults
  Interventions: Device: Measurement of brain activity (fNIRS, EEG)

INTERVENTIONS:
Device: Measurement of brain activity (fNIRS, EEG) — Brain activity assessments are conducted as a single session lasting approximately 60 minutes

SUMMARY:
The purpose of this study is to compare hemodynamic information from localized brain regions between stroke patients and healthy adults using brain activity data (fNIRS and EEG) and to assess the accuracy of early stroke diagnosis and classification predictions.

ELIGIBILITY:
Inclusion Criteria :

1. For Hemorrhagic Stroke Patients :

   * Adults aged between 19 and 80 years.
   * Diagnosed with hemorrhagic stroke through clinical observation and neuroimaging.
   * First-time hemorrhagic stroke patients.
   * Hemorrhagic stroke onset between 2 weeks and 12 months prior to screening.
   * Hemorrhagic lesion located in the cortex or subcortex.
   * Not taking medications that could affect brain hemodynamics, such as - antihypertensives, anticoagulants, antiplatelets, or antidepressants.
   * Able to read and understand the informed consent form and participate in questionnaires with sufficient language proficiency.
   * Voluntarily agree to participate in the study and provide written consent, with the ability to complete the study duration.
2. For Ischemic Stroke Patients :

   * Adults aged between 19 and 80 years.
   * Diagnosed with ischemic stroke through clinical observation and neuroimaging.
   * First-time ischemic stroke patients.
   * Ischemic stroke onset between 2 weeks and 12 months prior to screening.
   * Ischemic lesion located in the cortex or subcortex.
   * Not taking medications that could affect brain hemodynamics, such as antihypertensives, anticoagulants, antiplatelets, or antidepressants.
   * Able to read and understand the informed consent form and participate in questionnaires with sufficient language proficiency.
   * Voluntarily agree to participate in the study and provide written consent, with the ability to complete the study duration.
3. For Healthy Adults :

   * Adults aged between 19 and 80 years.
   * No history of stroke or transient ischemic attack (TIA).
   * No stroke risk factors such as hypertension, diabetes, or hyperlipidemia.
   * No chronic diseases (e.g., cardiovascular disease, chronic kidney disease, chronic lung disease).
   * No psychiatric conditions (e.g., depression, schizophrenia).
   * Not taking medications that could affect brain hemodynamics, such as antihypertensives, anticoagulants, antiplatelets, or antidepressants.
   * Able to read and understand the informed consent form and participate in questionnaires with sufficient language proficiency.
   * Voluntarily agree to participate in the study and provide written consent, with the ability to complete the study duration.

Exclusion Criteria :

* History of head trauma in the past 6 months.
* Ongoing severe chronic diseases (e.g., heart failure, chronic kidney disease, chronic lung disease).
* Severe psychiatric disorders such as schizophrenia, major depression, or bipolar disorder.
* Use of medications that could influence brain hemodynamics (e.g., antihypertensives, anticoagulants, antiplatelets, or antidepressants).
* Participation in a study and use of experimental drugs within the past 30 days.
* Pregnant or breastfeeding women.
* Major surgery in the past 6 months.
* Acute infections or inflammatory diseases.
* Cognitive impairment or dementia.
* Neurological disorders.
* Inability to understand the study procedures or unwillingness to provide voluntary consent.
* Any other clinical concerns deemed inappropriate for participation by the principal investigator or study team.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hemorrhagic stroke patients, ischemic stroke patients, and healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) signals | Brain activity assessments are conducted as a single session lasting approximately 60 minutes.
  Brainwaves are electrical currents generated when signals are transmitted between neurons in the nervous system. They vary depending on the mental and physical state of an individual and serve as one of the most critical indicators for measuring brain activity. Brainwaves can be recorded using devices such as electroencephalography (EEG), and in some cases, electrodes may be attached directly to the cortex. These devices are used to evaluate conditions such as brain damage, epilepsy, or other neurological disorders, as well as to legally determine brain death.

SECONDARY OUTCOMES:
Functional Near-Infrared Spectroscopy(fNIRS) signals | Brain activity assessments are conducted as a single session lasting approximately 60 minutes.
  The near-infrared spectrum between 800 nm and 2500 nm is commonly used to measure changes in reflectance, absorbance, and scattering coefficients associated with specific processes involving molecules or ions. This allows for the assessment of parameters such as oxygen saturation, blood flow, glucose levels, and energy metabolism in the bloodstream by analyzing changes in the distribution of oxyhemoglobin and deoxyhemoglobin in areas like the fingers, wrists, and brain blood flow. In this study, it is specifically utilized to measure oxygen saturation in brain blood flow.

IPD SHARING:
Plan to Share IPD: No